CLINICAL TRIAL: NCT04044105
Title: Impacting the Disposal of Unused Opioid Analgesics Through Education in the Orthopaedic Population: A Randomized Control Trial
Brief Title: Impacting the Disposal of Unused Opioid
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Craig J Della Valle, MD, Professor of Orthopaedic Surgery, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 18092505
Record Dates: First submitted 2019-08-01; First posted 2019-08-05 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Opioid Use and Disposal

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No Education (No Intervention): Patients in this arm receive no education regarding how to dispose of their opiate medication
- Pamphlet education (Experimental): Patients receive an educational pamphlet only, to be given at the preoperative teaching class, prior to their standard 3-week postoperative clinic appointment, and prior to their standard 6-week postoperative clinic appointment.
  Interventions: Other: Pamphlet education
- Pamphlet education + texts (Experimental): Patients receive an educational pamphlet, to be given at the preoperative teaching class, prior to their standard 3-week postoperative clinic appointment, and prior to their standard 6-week postoperative clinic appointment. In addition, 3 automated text messages sent at those same time points.
  Interventions: Other: Pamphlet education + texts

INTERVENTIONS:
Other: Pamphlet education — Patients receive an educational intervention explaining proper opioid disposal
  Arms: Pamphlet education
Other: Pamphlet education + texts — Patients receive an educational intervention and text message explaining proper opioid disposal
  Arms: Pamphlet education + texts

SUMMARY:
The purpose of this study is to compare the rates of proper opioid disposal in patients receiving an educational brochure compared to an automated text message delivered directly to patients' cell phones alongside the brochure, compared to no education on the subject.

DETAILED DESCRIPTION:
Opioids are used to treat acute pain after surgery, but can lead to misuse and abuse. Very few patients properly dispose of unused opioids and the majority of opioids are stored in the home in unlocked containers as opposed to being properly disposed of. Improper disposal of opioid medications is a concern due to the potential for nonmedical use and has the potential to cause injury or death for patients and their family members that can access the medications. The purpose of this study is to compare the rates of proper opioid disposal in patients receiving an educational brochure compared to an automated text message delivered directly to patients' cell phones alongside the brochure, compared to no education on the subject. There is evidence that an educational brochure significantly increases proper disposal rates, albeit only to about 25%. The goal of this study is to evaluate the impact of an educational pamphlet on proper opioid disposal in the total joint arthoplasty population, and to see if the addition of a text messaging system can increase further increase proper disposal rates.

ELIGIBILITY:
Inclusion Criteria:

* Any patient undergoing primary total hip or knee arthroplasty
* Age ≥18 years old

Exclusion Criteria:

* Patients allergic to oxycodone
* Patients consuming opioids during the 4 weeks prior to surgery
* Patients with a history of opioid dependence
* Patients undergoing revision total knee or hip arthroplasty
* Non-English speaking patients
* Age <18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 563 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-06-03 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Disposal rates | 6 weeks after surgery
  The rate of an arm's disposal is calculated by comparing the number that properly disposed of their excess medication to the number that did not

SECONDARY OUTCOMES:
Continued taking opiate rate | 6 weeks after surgery
  We will also look at whether the education affects the number of patients that continue taking opiates

CONTACTS AND LOCATIONS:
Overall Officials: Craig Della Valle, MD, Principal Investigator — Rush
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No